CLINICAL TRIAL: NCT05919121
Title: Effect Of Hydrocortisone Phonophoresis Versus Iontophoresis In Patients With Subacromial Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohsen Ibrahim, Principal Investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOHSEN_IBRAHIM_phd
Record Dates: First submitted 2023-06-14; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Impingement Syndrome; Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic exercise group (Active Comparator): Therapeutic exercise group, group A.
  Interventions: Other: Therapeutic exercise
- hydrocortisone phonophoresis group (Experimental): This group (B) will receive the same exercise program in addition to hydrocortisone phonophoresis. Patients will receive topical medium phonophoresis of 10% hydrocortisone gel.
  Interventions: Other: Therapeutic exercise; Other: hydrocortisone phonophoresis
- hydrocortisone iontophoresis group (Experimental): This group (C) will receive the same exercise program in addition to hydrocortisone iontophoresis.
  Interventions: Other: Therapeutic exercise; Other: hydrocortisone iontophoresis

INTERVENTIONS:
Other: Therapeutic exercise — 1. Stretching exercise of posterior shoulder capsule
  2. Strengthening exercises: consists of 6 strengthening exercises all of which have been recommended as essential for any shoulder rehabilitation program.
  3. The remaining 2 exercises are the seated press-up and the elbow push up. Both will be performed to fatigue or for a maximum of 25 repetitions. The quality of all repetitions of each exercise will continuously monitored by the investigator of the study
Other: hydrocortisone phonophoresis — In this study, the effective area of radiation (ERA) in the mode continuous (100 percent) is 5 cm2, in 1 MHz and 0.7 W/cm2, with four ERA treated areas. Therapy lasted five minutes (three minutes in the insertion of the supraspinatus and 37 two minutes in the infraspinatus insertion) three times weekly over 6 weeks in addition to therapeutic exercises
  Arms: hydrocortisone phonophoresis group
Other: hydrocortisone iontophoresis — A direct current electrical stimulation unit will be used to apply iontophoresis. The unit has two electrodes; one electrode is for the negative current, and one is for the positive current. The Active (Negative) electrode will be placed on the anterolateral aspect of the shoulder joint. The passive electrode: will be placed on the upper arm region. Intensity of the current: Between the range of 3-5 mA at the point of sensation of patient was set. Treatment duration: Calculated accordingly with intensity of current. Method of application: hydrocortisone gel 10% will be administered by applying on the active rubber electrode for each session three times weekly over 6 weeks in addition to therapeutic exercises.
  Arms: hydrocortisone iontophoresis group

SUMMARY:
The purpose of this study will be to compare the efficacy of adding hydrocortisone phonophoresis or iontophoresis on pain, function, range of motion and shoulder external rotation isometric strength in patients with subacromial impingement syndrome.

DETAILED DESCRIPTION:
Routine physiotherapy has been advocated was an effective treatment for SIS. However, there is lack of best exercise treatment and lots of studies are under consideration. According to published data focused on management of shoulder pain, it looks like that therapeutic exercise is not sufficient to treat SIS and it is compulsory to combine with other remedies to get the best results

ELIGIBILITY:
Inclusion Criteria:

1. All patients were diagnosed as unilateral SIS with stage II Neer classification > 3 months.
2. Positive impingement sign (Neer's test or Hawkins-Kennedy test), / painful arc during active arm elevation, pain or weakness with resisted isometric external rotation or resisted scapular plane abduction with the humeral internal rotation (empty can test)
3. The age of patients ranged from 18 - 60 years old.
4. Both genders will be involved.
5. Shoulder pain scores more than 5 on a numeric rate scale for pain of 0- 10.
6. Failure to respond to conservative NSAID.

Exclusion Criteria:

1. Frozen shoulders.
2. Arthritis of the shoulder.
3. Shoulder instability.
4. Pregnant women.
5. A pacemaker.
6. Previous shoulder surgery.
7. History of dislocation of the shoulder.
8. Internal metallic fixation.
9. Malignancy.
10. Previous corticosteroid injection.
11. Rheumatoid arthritis
12. Partial or Full thickness tear of the rotator cuff.
13. Cervical radiculopathy.
14. Physiotherapeutic shoulder treatment within the last 3 months.
15. The patients will randomly be assigned into 3 equal groups, 20 patients for each group.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in isometric shoulder strength | at baseline and after 6 weeks of intervention
  A handheld Lafayette dynamometer will be used to evaluate the peak shoulder External Rotation muscles isometric strength
Assessing the change in Shoulder Pain and Disability | at baseline and after 6 weeks of intervention
  By using Shoulder Pain and Disability Index (SPADI). SPADI has been found to be the quickest (within five minutes) and easiest to complete, as well as being more responsive to change. The SPADI is considered to be, by comparison, one of the most useful instruments about the shoulder joint, and has been tested in various clinical settings. The SPADI is a 13-item shoulder function index on the ability of responders to carry out basic activities of daily living. Each item is scored by a numeric rating scale that ranges from 0 (no pain/no difficulty) to 10 (worst pain imaginable/so difficult it required help).
Assessing the change in shoulder Range Of Motion | at baseline and after 6 weeks of intervention
  In this study shoulder ROM will be measured by using Electrogoniometer (flexion, abduction and internal rotation ranges will be measured in degrees), which eliminates the need to manually score each measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Ibrahim, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic faculty of physical therapy, horus university, egypt, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided